CLINICAL TRIAL: NCT03038191
Title: Epi-collect: Data Collection During Video EEG Monitoring and at Patient's Home
Status: Terminated | Type: Observational
Why Stopped: Sponsor stopped funding
Sponsor: Medial Research Ltd. (Industry)
Responsible Party: Principal Investigator, Firas Fahoum, MD, Director, Epilepsy and EEG Service Neurology Division, Tel-Aviv Sourasky Medical Center
Other Study IDs: CA-EPIPRO-TASMC-HOSP-02
Record Dates: First submitted 2017-01-12; First posted 2017-01-31 (Estimated); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Neuroelectrics Enobio 8(R) — Monitoring

SUMMARY:
Epilepsy is a group of neurological disorders characterized by propensity for spontaneous epileptic seizures. Epileptic seizures are the result of excessive and abnormal nerve cell activity in the brain. About 0.7-1% of the world population suffers from seizures. The most common treatment is based on seizure medications that enables about 2/3 of the patients to control their seizures. However, about 20 million patients worldwide, suffer from unpredictable seizures without remedy, and are resistant to medication.

In this study EEG and other physiologic signals are collected using wearable sensors, from Epilepsy patients who are at risk of experiencing seizures. The collected signals will be used for developing algorithms that may identify pre-seizure and seizure related periods.

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* Known diagnosis of Epilepsy
* Expected to experience seizures during the period of the study as determined by the PI.
* Able to meet with the Sponsor representative at home

Exclusion Criteria:

* Trauma/broken skin on forehead.
* Patient can not follow or comply with instructions
* Patients who are unable to independently provide an informed consent
* Patients with major psychiatric co-morbidities
* Patients with psychogenic non-epileptic seizures

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult epilepsy patients who are admitted to the video EEG unit and are expected to experience seizures during hospitalization
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2017-03-08 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Successful data collection during hospitalization | 12 hours daily for up to 5 days
  Continuous recording from wearable sensors of physiologic signals during hospitalization in the video EEG unit
Successful data collection during at home monitoring | 12 hours daily for up to 14 days
  Continuous recording from wearable sensors of physiologic signals during at home monitoring

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No